CLINICAL TRIAL: NCT02612714
Title: Statin Therapy is Associated With Low Testosterone and Sexual Function in Men With Type 2 Diabetes
Brief Title: Statin Lowering Testosterone and Sexual Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ching Jung Hsieh, Chief of General Internal Medicine, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 103-2005C
Record Dates: First submitted 2015-11-07; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Sexual Dysfunction
Keywords: diabetes; hypercholesterolemia; sexual dysfunction; statin; testosterone
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Diabetes Mellitus; Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- medication status (Other): Rosuvastatin 5 mg qd for 6 months, Quitted rosuvastatin for 6 months, Re-administrated rosuvastatin for 6 months
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — All parameters were measured before statin treatment, after 6 months of statin treatment and 6 months after discontinuing statin treatment. Scores of the sexual health inventory for men (SHIM) were also evaluated.
  Other Names: Cresto

SUMMARY:
Statins may decrease serum testosterone levels via decreasing cholesterol. This longitudinal study detected the effects of rosuvastatin on free testosterone levels and sexual function in men with type 2 diabetes.

Methods:

Investigator enroll 150 men with type 2 diabetes and hypercholesterolemia. Biochemical assessments include serum total cholesterol (TC), low-density lipoprotein (LDL), high-density lipoprotein, triglyceride, prolactin, thyroid-stimulating hormone, luteinizing hormone, follicle stimulating hormone, total testosterone and serum sex hormone binding globulin (SHBG). All parameters are measured before statin treatment, after 6 months of statin treatment and 6 months after discontinuing statin treatment. Scores of the sexual health inventory for men (SHIM) are also evaluated.

DETAILED DESCRIPTION:
Autonomic neuropathy and hypogonadism are the cause of impotence in men with diabetes. Hypercholesterolemia is also one of the dominant co-morbidity of diabetes. Many men with diabetes are being treated with statins to low down the serum levels of cholesterol. However, cholesterol is the major substrate for testosterone biosynthesis, statin may decrease serum testosterone levels via decreasing cholesterol level. In previous studies, few longitudinal studies with few enrolled subject were done before and with conflict results. Free testosterone is also not routinely used, so compromised the accuracy. The investigators will analyze the effect of statins on free testosterone levels in a longitudinal study of men with type 2 diabetes and do animal study to realize if the statin will influence the sex organ of rat.

Methods:

Investigator will enroll 150 men with type 2 diabetes and hypercholesterolemia. Clinical and biochemical assessments include blood pressure, HbA1C, lipid profile, height, weight, and waist circumference, luteinizing hormone (LH), follicle stimulating hormone (FSH) and free testosterone , which will be measured before statin treatment, after 3 months of statin treatment and then after quitted statin treatment for 3 months, and also give questionnaire about sex function.

The investigators expect:

1. Statin may potentially lead to hypogonadism or impotence In men with type 2 diabetes.
2. The relationship between blood glucose, lipid profile, blood pressure, anthropometric measures and serum free testosterone levels may also be revealed.
3. If this hypothesis is adverse, statin treatment will not influence gonadal function and has that side effect.

ELIGIBILITY:
Inclusion Criteria:

1. Type2 diabetes mellitus for more than 2 year.
2. Male subjects
3. Not received statin therapy for more than 1 year
4. Normal sexual activity
5. No hypogonadism history.

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Duration of diabetes less than 2 years and more than 10 years
3. Renal function impairment (creatinine level > 1.4 mg/dl)
4. Cancer or organic disease associated with hypogonadism,
5. With testosterone on antiandrogen drug therapy

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
serum testosterone | up to 24 weeks
  The measure is a composite outcome measure consisting of multiple measures. Serum testosterone measured after 24 weeks statin treatment, after quitted statin for 24 weeks and after 24 weeks of re-administrating statin

SECONDARY OUTCOMES:
sexual function evaluation | up to 24 weeks
  The measure is a composite outcome measure consisting of multiple measures. Sexual function measured by questionaire after 24 weeks of statin treatment, after quitted statin for 24 weeks and after 24 weeks of re-administrating statin

CONTACTS AND LOCATIONS:
Overall Officials: Ching Jung Hsieh, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung, Kaohsiung City, Kaohsiung, Taiwan